CLINICAL TRIAL: NCT03330041
Title: Aesthetic Outcome of Running Cuticular Suture Distance (2mm vs 5mm) From Wound Edge on the Closure of Linear Wounds on the Head and Neck: a Randomized Evaluator Blinded Split Wound Comparative Effective Trial.
Brief Title: Suturing Distance From the Wound Edge, 2 mm vs 5 mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1115596
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Cutaneous Sutures and Scar Cosmesis
Keywords: Cutaneous Sutures; Scar Cosmesis; Linear Wound Closure; Wound Cosmesis

STUDY DESIGN:
Intervention Model Description: At the follow-up visit, two blinded observers will record their scores independently using the physician observer scar assessment score instrument (POSAS).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fast absorbing gut suture placed 2 mm apart (Experimental): Wound closed with sutures spaced 2 millimeters apart will be treated in a simple, interrupted cutaneous suture pattern
  Interventions: Device: Fast absorbing gut suture
- Fast absorbing gut suture placed 5 mm apart (Experimental): Wound closed with sutures spaced 5 millimeters apart will be treated in a simple, interrupted cutaneous suture pattern
  Interventions: Device: Fast absorbing gut suture

INTERVENTIONS:
Device: Fast absorbing gut suture — Fast absorbing surgical gut suture is a strand of collagenous material

SUMMARY:
This study aims to investigate whether the spacing of the interrupted cutaneous sutures affects surgical wound cosmesis on the face and neck. In other words, the investigators would like to determine which of the following yields a more cosmetically appealing scar: many closely approximated sutures or fewer, more widely spaced sutures. The investigators wish to compare the effects of two versus five millimeter spacing between sutures.

DETAILED DESCRIPTION:
Sutures are the standard of care in repairing cutaneous wounds. The majority of surgical reconstructions following a Mohs micrographic surgery and standard surgical excisions require two layers of sutures: a deep (subcutaneous) layer and a top (cutaneous) layer. The deep layer dissolves naturally whereas the top layer may necessitate removal if non-absorbable sutures are used. This study aims to investigate whether the spacing of the interrupted cutaneous sutures affects surgical wound cosmesis on the face and neck. In other words, the investigators would like to determine which of the following yields a more cosmetically appealing scar: many closely approximated sutures or fewer, more widely spaced sutures. The investigators wish to compare the effects of two versus five millimeter spacing between sutures. It is possible that fewer, more widely spaced sutures may leave more open space in the wound, leaving more tension to pull on those few sutures, possibly encouraging the wound to dehisce and make it harder to approximate the wound edges yielding a less cosmetically appealing scar compared to placing many closely approximated sutures which would decrease the tension and likely better approximate the wound edges yielding a more cosmetically appealing scar. On the other hand, the investigators may find that suture spacing has no effect on wound cosmesis and that placing fewer, more widely spaced sutures is much more time efficient. The investigators may also find that the effect of suture spacing on wound cosmesis is dependent on wound tension. For example, perhaps the suture pacing would have no effect on the cosmesis of a wound under no tension, however, for a wound under high tension, it is possible that many closely approximated sutures would yield better cosmetic results for the reasons listed above.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the trunk and extremities with predicted primary closure
* Willing to return for follow up visit.

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 4 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sklar LR, Pourang A, Armstrong AW, Dhaliwal SK, Sivamani RK, Eisen DB. Comparison of Running Cutaneous Suture Spacing During Linear Wound Closures and the Effect on Wound Cosmesis of the Face and Neck: A Randomized Clinical Trial. JAMA Dermatol. 2019 Mar 1;155(3):321-326. doi: 10.1001/jamadermatol.2018.5057. PMID 30649154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized clinical trial was conducted at the University of California, Davis dermatology clinic from November 28, 2017, to June 15, 2018.
Groups:
- All Participants: A split wound model was used, where half of the wound was repaired with sutures placed 2 millimeters apart and the other half is repaired with sutures placed 5 millimeters apart. A predetermined, concealed randomization number was obtained from the RedCap randomization module, which specified how Side A was treated. Side B was treated the opposite way as A.
Period: Overall Study
Arm/Group | All Participants
Started | 50
Completed | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Fast Absorbing Gut Suture Placed 2 mm and 5 Mmapart: Wound closed with sutures spaced 2 and 5 millimeters apart will be treated in a simple, interrupted cutaneous suture pattern
  Fast absorbing gut suture: Fast absorbing surgical gut suture is a strand of collagenous material
Arm/Group | Fast Absorbing Gut Suture Placed 2 mm and 5 Mmapart
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Patient Posas Score
Description: Scale name: Patient Observer Scar Assessment Score. Scale measures six parameters of scars, each using a 10-point scoring system (the six categories are summed to achieve the POSAS score - totals range from 6 to 60), with 1 representing normal skin & 10 representing the most severe scar imaginable.
Time Frame: 3 months following procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fast Absorbing Gut Suture Placed 2 mm Apart: Wound closed with sutures spaced 2 millimeters apart will be treated in a simple, running cuticular suture pattern.
  Fast absorbing gut suture: Fast absorbing surgical gut suture is a strand of collagenous material.
- Fast Absorbing Gut Suture Placed 5 mm Apart: Wound closed with sutures spaced 5 millimeters apart will be treated in a simple, running cuticular suture pattern.
  Fast absorbing gut suture: Fast absorbing surgical gut suture is a strand of collagenous material.
Arm/Group | Fast Absorbing Gut Suture Placed 2 mm Apart | Fast Absorbing Gut Suture Placed 5 mm Apart
Number analyzed (Participants) | 48 | 48
score on a scale | 10.2 (4.7) | 11.5 (6.4)

2. Secondary Outcome: Width of Scar
Description: A secondary endpoint will include the width of the scar 1 cm from midline on each side.
  This measurement will be reported in mm
Time Frame: 3 months following procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fast Absorbing Gut Suture Placed 2 mm Apart | Fast Absorbing Gut Suture Placed 5 mm Apart
Number analyzed (Participants) | 48 | 48
mm | 0.9 (0.6) | 0.8 (0.4)

3. Secondary Outcome: Erythema
Description: If one half of the scar has more associated erythema, this will be noted number of people with erythema after treatment will be reported
Time Frame: 3 months following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fast Absorbing Gut Suture Placed 2 mm Apart | Fast Absorbing Gut Suture Placed 5 mm Apart
Number analyzed (Participants) | 48 | 48
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: At 3-Month Follow-up
Arm/Group | Fast Absorbing Gut Suture Placed 2 mm Apart | Fast Absorbing Gut Suture Placed 5 mm Apart
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03330041/Prot_SAP_000.pdf